CLINICAL TRIAL: NCT05855122
Title: Study of Safety and ASCT-related Symptom Burden Optimization of Tocilizumab in ASCT Following High-dose Melphalan Conditioning in Patients With Multiple Myeloma
Brief Title: Safety and ASCT-related Symptom Burden Optimization of Tocilizumab in ASCT Following HD Melphalan Conditioning for Multiple Myeloma Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Fu chengcheng PhD, Principal Investigator, The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Tocilizumab-ASCT-MM08
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab (Experimental)
  Interventions: Drug: Tocilizumab
- no-Tocilizumab (No Intervention)

INTERVENTIONS:
Drug: Tocilizumab — Pateients enrolled in Tocilizumab group will receive tocilizumab(8mg/kg) at day -7 before transfusion of stem cells.
  Arms: Tocilizumab

SUMMARY:
Background: Autologous hematopoietic stem cell transplantation(ASCT) is an important part treatment for patients with multiple myeloma. Retrospective analysis from our center showed that incidence of oral mucositis and gastrointestinal symptoms was higher during ASCT for melphalan as conditioning regimen in patients with multiple myeloma. Objective: Safety and optimization of ASCT-related symptom burden of tocilizumab for melphalan as a conditioning regimen in ASCT for multiple myeloma is explored. Methods: The patient who is enrolled will be randomly divided into two groups in a proportion of 1:1 to respectively receive tocilizumab(8mg/kg) at day -7 before transfusion of stem cells or not. There will be enroll 48 patients according to inclusion and exclusion criteria totally. Adverse events and MDASI score during ASCT between two groups will be recorded and analyzed. Primary endpoint: MDASI, Security; Secondary endpoints: time to neutrophil engraftment; time of platelet implantation; efficacy (ORR) after autologous hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with multiple myeloma eligible for autologous hematopoietic stem cell transplantation;
2. Secretory MM should have measurable markers, including:

   1. specific M protein value (≥5g/L)；
   2. and/or involved flc ≥100mg/L；
   3. and/or measurable extramedullary foci (diameter>1cm on CT);
3. Age ≥ 18 years and ≤ 70 years, male or female;
4. PR and above are obtained after induction therapy according to the IMWG response criteria;
5. Mononuclear cells ≥2×10^8/kg body weight, CD34+ cells≥2×10^6/kg body weight;
6. ECOG 0-2, with life expectance ≥3 months;
7. ALT/AST level ≤2.5 times of the maximum of normal range; total bilirubin≤2 times of normal maximum；
8. Neutrophil count≥ 1.5×10^9/L, platelet count ≥50×10^9/L;
9. Normal Left ventricular ejection fraction , NYHA stage 1, lung function GOLD stage 1;
10. Willing to accept the possibility of potential adverse events and efficacy observation by the investigators;
11. Being able to understand and signing the written consent, which should be signed prior to any procedure of the trial.

Exclusion Criteria:

1. With ≥2 degree of peripheral neuropath or with pain;
2. Having received any of the medicine of the experiment regimen within 30 days prior to enrollment, pain-relieving radiotherapy is allowed;
3. With severe pulmonary/cardiac disfunction (including history of QT interval elongation, ventricular tachycardia, ventricular fibrillation, myocardial infraction) or other severe organ malfunction;
4. Patients in pregnancy or lactation;
5. Allergic constitution or being allergic to any drug within the regimen of the trial;
6. With uncontrolled mental diseases;
7. With active infection;
8. With active hepatitis;
9. HIV positive;
10. History of other malignant tumor within 5 years prior to enrollment; except for the case of in situ cervical cancer and non-malignant melanoma;
11. With other conditions that the investigators think unfit for the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
MDASI questionnaire | day -7~day 100 after stem cells transfusion
  MDASI, also as the M. D. Anderson Symptom Inventory, is a brief measure of the severity and impact of cancer related symptoms. Each symptom is rated on an 11-point scale (0 -10) to indicate the presence and severity of the symptom, with 0 meaning "not present" and 10 meaning "as bad as you can imagine." Each symptom is rated at its worst in the last 24 hours.
Adverse events | day -7~day 100 after stem cells transfusion
  recording adverse events according to CTCAE5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No